CLINICAL TRIAL: NCT05324371
Title: A Pilot Study to Assess WATCHMAN FLX™ Implants by Cardiac Computed Tomography, Magnetic Resonance Imaging and Transesophageal Echocardiography: WATCHMAN FLX™ CT
Brief Title: WATCHMAN FLX™ CT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2423
Record Dates: First submitted 2022-03-17; First posted 2022-04-12 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: The Focus of the Study is to Reduce the Risk of Stroke and Life-threatening Bleeding Events in Patients With Non-valvular Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Arm (Experimental): WATCHMAN FLX™ device implantation
  Interventions: Device: Watchman FLX Device

INTERVENTIONS:
Device: Watchman FLX Device — Left atrial appendage closure using the Watchman FLX device

SUMMARY:
WATCHMAN FLX™ CT is a prospective, single-arm, single-center, post-market investigation to assess device tissue coverage in subjects with non-valvular atrial fibrillation (AF) who receive the WATCHMAN FLX device to reduce the risk of stroke. Serial advanced imaging modalities such as CT and TEE will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of legal age to participate in the study per the laws of their respective geography.
* Subject has documented non-valvular atrial fibrillation (i.e., atrial fibrillation in the absence of moderate or greater mitral stenosis or a mechanical heart valve).
* Subject is clinically indicated for a WATCHMAN FLX device.
* Subject is deemed suitable for the protocol-defined pharmacologic regimen.
* Subject or legal representative is able to understand and willing to provide written informed consent to participate in the study.
* Subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

* Subject is currently enrolled in another investigational study, except if the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatment.
* Subject has eGFR <30 mL/min (chronic kidney disease stage IV or stage V).
* Subject is contraindicated for TEE.
* Subject requires long-term anticoagulation therapy for reasons other than AF-related stroke risk reduction (e.g., due to an underlying hypercoagulable state).
* Subject had or is planning to have any cardiac or non-cardiac intervention or surgical procedure within 30 days prior to or 60 days after implant (including, but not limited to, cardioversion, percutaneous coronary intervention, cardiac ablation, cataract surgery, etc.).
* Subject had a prior stroke (of any cause, whether ischemic or hemorrhagic) or transient ischemic attack (TIA) within the 30 days prior to enrollment.
* Subject had a prior major bleeding event per ISTH definitions within the 30 days prior to enrollment. Lack of resolution of related clinical sequelae or planned and pending interventions to resolve bleeding/bleeding source are a further exclusion regardless of timing of the bleeding event.
* Subject has an active bleed.
* Subject has a reversible cause for AF or has transient AF.
* Subject has no LAA or the LAA is surgically ligated.
* Subject has had a myocardial infarction (MI) documented in the clinical record as either a non-ST elevation MI (NSTEMI) or as an ST-elevation MI (STEMI), with or without intervention, within 30 days prior to enrollment.
* Subject has a history of atrial septal repair or has an atrial septal defect/patent foramen ovale (ASD/PFO) device.
* Subject has a known contraindication to percutaneous catheterization procedure.
* Subject has a cardiac tumor.
* Subject has signs/symptoms of acute or chronic pericarditis.
* Subject has an active infection.
* There is evidence of tamponade physiology.
* Subject has New York Heart Association Class IV congestive heart failure at the time of enrollment.
* Subject is of childbearing potential and is, or plans to become, pregnant during the time of the study (method of assessment per study physician's discretion).
* Subject has a documented life expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Erik Nielsen-Kudsk, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device Arm
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Device Arm: WATCHMAN FLX Device Implantation
Arm/Group | Device Arm
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Hypoattenuated Thickening (HAT) on the Surface of the Device
Description: Serial measurement of any HAT on the surface of the device at 14 days, 45 days and 3 months post implant as assessed by core lab using CT imaging
Time Frame: 14 days to 3 months post implant
Measure: Count of Participants; unit: Participants
Groups:
- 14 Days: WATCHMAN FLX™ 14 days post device implantation
- 45 Days: WATCHMAN FLX™ 45 days post device implantation
- 3 Months: WATCHMAN FLX™ 3 months post device implantation
Arm/Group | 14 Days | 45 Days | 3 Months
Number analyzed (Participants) | 24 | 23 | 23
Participants | 5 | 3 | 2

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Site Reported
Arm/Group | Device Arm
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Arm (N=25)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (3)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Graft Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Arm (N=25)
Device Related Thrombosis (General disorders) | 2 (2)
Catheter Site Haemorrhage (General disorders) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05324371/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05324371/SAP_001.pdf